CLINICAL TRIAL: NCT06275737
Title: Trimodal Peri Operative Prehabilitation for Upper Oesogastric and Pancreatic Cancer: A Multicenter, Two-cohort, Open-label, Single-arm POP-UP GERCOR Study
Brief Title: POP-UP: a Single-arm, Two-cohort Study: Trimodal Prehab for Upper GI and Pancreatic Cancer
Acronym: POP-UP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: POP-UP G-128
Record Dates: First submitted 2024-02-01; First posted 2024-02-23 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: Two-cohort, open-label, single-arm feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 and Cohort 2 (Other): Cohort 1 - Patients with PDAC
  Cohort 2 - Patients with OGC
  Interventions: Other: Prehabilitation program

INTERVENTIONS:
Other: Prehabilitation program — Cohort 1 - Prehabilitation program will be implemented during the last cycles of neoadjuvant chemotherapy (cycle 5 - cycle 6 or cycle 6 - cycle 8) and the weeks preceding surgery (planned 3-4 weeks after the last chemotherapy cycle)
  Cohort 2 - Prehabilitation program will be implemented during the last cycles of neoadjuvant chemotherapy (cycle 2 - cycle 4) and the weeks preceding surgery (planned 3-4 weeks after the last chemotherapy cycle)

SUMMARY:
This is a multicenter, two-cohort, open-label, single-arm feasibility study. The primary objective is to assess the feasibility of the 8-week trimodal prehabilitation program alongside perioperative triplet chemotherapy in eligible patients with localized pancreatic ductal adenocarcinoma (PDAC) or oesogastric cancer (OGC) .

DETAILED DESCRIPTION:
The POP-UP study aims to evaluate the feasibility and preliminary efficacy of an 8-week trimodal pre/posthabilitation program (consisting of personalized Adapted Physical Activity [APA], nutritional assessment, and psychological support) with remote monitoring of the APA sessions and nurse coordination in patients with localized (resectable or borderline resectable) PDAC who are treated with neoadjuvant or induction treatment (FOLFIRINOX: 5-fluorouracil/folinic acid, oxaliplatin, irinotecan) prior to surgery and with resectable OGC treated with perioperative chemotherapy (FLOT: 5-fluorouracil/folinic acid, oxaliplatin, docetaxel).

The prehabilitation program will be conducted during neoadjuvant chemotherapy and the 3-5 weeks prior to surgery for a total of 8 weeks before surgery. There will be a total of three prehabilitation hospital days during the prehabilitation program.

The preoperative prehabilitation will include:

* Once per month, a prehabilitation hospital-day with functional capacities assessment with validated tests made by a physiotherapist or an APA professional (according of center resources/functioning), medical and nurse assessment evaluating performance status, chemotherapy toxicity and tolerance, and nutritional assessment (according to the functioning of each center it will be made by these professionals -with university training on nutrition- or a dietician). A therapeutic training session on the adherence to the prehabilitation program will be done by the nurse (trained in therapeutic education).
* Weekly, an APA professional trainer will follow via using app (Activiti®) the APA home-based program. It will be based on the functional capacities assessment made during the prehabilitation hospital day. The exercise training program will consist of twice per week autonomy sessions, supervised and adapted by the APA professional, and once per week a guided session with the APA professional. The patient will have a total of 3 physical activity sessions per week.
* Once per week, the nurse practitioner (or case manager, according to center functioning) will evaluate the patient via a videoconference to assess the chemotherapy toxicity and tolerance and patient's weight modifications.

The posthabilitation program will start for a total of 8 weeks, one week after surgery discharge. The structure is the same as the prehabilitation program except for the follow of chemotherapy toxicity and tolerance that will be replaced by the follow of the surgical complications/consequences.

There will be a total of three posthabilitation days at hospital during the posthabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated patient informed consent form (ICF) and willingness to comply with all study procedures and availability for the study duration,
* Histologically or cytologically localized PDAC or OGC validated by the multidisciplinary team,
* Indication to a preoperative treatment withtriplet chemotherapy for ≥ 4 cycles (8 weeks), Note: Patient treated for PDAC, first cycle without oxaliplatin is authorized.
* Age > 18 years; If aged ≥ 75 years: G8 score must be ≥ 14 and if < 14 validation of oncogeriatric specialist,
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-1 at inclusion visit (first prehabilitation hospital-day),
* No prior treatment for PDAC or OGC before screening visit,
* At least one measurable or evaluable lesion as assessed by Computerized Tomography scan or Magnetic resonance imaging according to RECIST 1.1 and feasibility of repeated radiological assessments on baseline imaging before starting chemotherapy,
* Adequate hematologic and end-organ function allowing the triple combination chemotherapy protocol,
* Registration in a national health care system (PUMa - Protection Universelle Maladie included).

Exclusion Criteria:

* Evidence of metastatic disease at imaging (validated in multidisciplinary team evaluation),
* Histology of other than adenocarcinoma,
* Any medical (including cardiovascular, respiratory, psychiatric, musculoskeletal, or neurological) condition contra-indicating exercise practice,
* Patients with medical contraindication to surgery due to general condition or comorbidities
* Pregnancy or breast-feeding,
* Patient under a legal protection regime (guardianship, curatorship, judicial safeguard) or administrative decision or incapable of giving his/her consent,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with successful completion of an 8-week trimodal prehabilitation program | 8 weeks
  The success of prehabilitation is defined by the achievement of the following three criteria:
  1. Completion of at least 75% of the planned APA sessions: 6 of 8 sessions with an APA professional and 12 of 16 sessions in autonomy with remote APA supervision and
  2. Completion of at least 75% of the nutritional evaluations: 6 of 8 planned evaluations and
  3. Psychological or psychiatric visit before the surgery in function of practice center /resources if a psychological need is shown by Hospital Anxiety and Depression Scale

SECONDARY OUTCOMES:
Success rate (as defined above) for Adapted Physical Activity (APA), nutritional, and psychological interventions measured separately. | 8 weeks
  The success of APA, nutritional, and psychological interventions analyzed separately
Health-related quality of life (HRQoL) assessment | Up to 3 years
  HRQoL assessed using the EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) questionnaire for all patients.
Rate of patients who start and complete post-habilitation Adapted Physical Activity (APA) sessions | 8 weeks
  Rate of patients who start and complete post-habilitation APA sessions; reasons for drop-out.
Nutritional status assessment | 8 weeks
  Nutritional status assessment by:
  Body mass index (BMI) - BMI will be calculated by dividing mass in kilograms (kg) by height in meters squared (m2).
  Food intake will be measured by visual analog scale SEFI [Score d'Evaluation Facile des Ingesta=Ingesta Easy Evaluation Score]). The SEFI is a score rated from 0 (nothing is consumed) to 10 (everything is consumed) in whole numbers. A SEFI < 7/10 corresponds to decreased food intake and is associated with risk of malnutrition. A SEFI ≥ 7 corresponds to satisfactory food intake.
Physical/functional test assessment | 8 weeks
  Functional tests: 6-minute waking test, handgrip test, one minute sit-to-stand (STS), assessment of Borg scale post physical exercise will be measured.
  A 6-minutes walking test (distance measured in meters) will be performed. Dyspnea will be measured by the Borg scale Borg scale (ratings of the effort to breathe; a scale from 0 to 10, where 0 represents no dyspnea and 10 represents maximal dyspnea). Scores are obtained at the end of the walking test and reflect the maximum degree of dyspnea at any time during the walk test.
  Handgrip test - hand grip strength will be measured using dynamometer in sitting position and will be expressed in kilograms (kg).
  One-minute sit-and-stand test - Patients will perform stand-and-sit transitions on the chair as many times as possible within one minute. Number of of repetitions will be measured.
Number of patients with reduced chemotherapy tolerance | 8 weeks
  Chemotherapy tolerance: toxicities (Common Terminology Criteria for Adverse Events [CTCAE] v5.0) of grade ≥ 3, toxicities requiring hospitalization, treatment delays or dose reduction due to toxicities
Number of patients with chemotherapy dose modification | 8 weeks
  Modification of the chemotherapy related dose-intensity relation on the completion or not of the prehabilitation program
Rate of patients who complete the strategy | 8 weeks
  Rate of patients who undergo surgery and the total number of planned perioperative chemotherapy cycles, and number of cycles received / number of cycles planned
Number of patients with Granulocyte-colony stimulating factor (G-CSF) prescription and grade ≥ 2 neutropenia | 8 weeks
  rate of patients' with GCSF prescription and grade ≥ 2 neutropenia
Rate of patients with exocrine pancreatic insufficiency and the dose of pancreatic enzyme consumption | 8 weeks
  Preoperative and post-operative fecal elastase and pancreatic enzymes prescription and reported consumption
Rate of surgical complications | At 30 days after surgery
  Rate of surgical complications requiring reintervention or rehospitalisation (grade ≥ 3 in Clavien-Dindo classification) within 90 days after surgery, length of hospital stay
Overall survival (OS) assessment | From inclusion up to 12 months after surgery
  OS defined as time between the date of inclusion and 12 months after surgery
Disease-free survival (DFS) assessment | From inclusion up to 12 months after surgery
  DFS defined as the time between the date inclusion and the date corresponding at 12 months after surgery
Adherence to Adapted Physical Activity (APA) program assessment | 8 weeks
  Adherence to the APA program: by patient reported outcomes collected via Activiti® app and the APA professional assessment
Physical activity behavior changes assessment | 8 weeks
  Simplified International Physical Activity Questionnaire (IPAQ-S) will be administrated to assess physical activity and sedentary behavior changes.
  It is a 7-item questionnaire in which duration (hours and minutes per day), frequency (times per week), and intensity (walking, moderate and vigorous) of the previous 7 days will be collected. Sedentary time (self-reported time spent sitting) in the same time period will be recorded (hours/min/day).
Nurse coordination | 8 weeks
  Nurses will evaluate chemotherapy tolerance with the CTCAE V5.0 (Grade ≥ 3) and weight lose once per week with Activiti® application.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Neuzillet, MD, Principal Investigator — Institut Curie, Saint-Cloud
Locations (4):
- France (4):
  - Centre Hospitalier Universitaire de Lille, Lille
  - Institut Paoli Calmettes, Marseille
  - Institut Curie, Saint-Cloud
  - Institut de Cancerologie de L'Ouest Rene Gauducheau, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No